CLINICAL TRIAL: NCT02337660
Title: Involvement of Steatosis-induced Glucagon Resistance in Hyperglucagonaemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: The Novo Nordisk Foundation Center for Basic Metabolic Research (Other)
Responsible Party: Principal Investigator, Malte Palm Suppli, Research year assistant, University Hospital, Gentofte, Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SIRG-1
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy, lean (Experimental): 15 healthy, lean subjects.
  Will have a liver biopsy, and on the experimental day a pancreatic clamp will be performed.
  Interventions: Procedure: Liver biopsy; Other: Pancreatic clamp
- Obese, otherwise healthy (Experimental): 15 obese, otherwise healthy subjects
  Will have a liver biopsy, and on the experimental day a pancreatic clamp will be performed.
  Interventions: Procedure: Liver biopsy; Other: Pancreatic clamp

INTERVENTIONS:
Procedure: Liver biopsy — One ultrasound guided liver biopsy
Other: Pancreatic clamp — I.v. infusions of somatostatin and insulin (basal rate) for will be adminstered for 3 hours. Glucagon will administered for 3 hours in total with infusion rates at a basal and a high physiological rate for 1.5 hours each.

SUMMARY:
The purpose of this study is to examine whether non-alcoholic fatty liver disease (NAFLD) is associated with hepatic glucagon resistance and hyperglucagonemia.

DETAILED DESCRIPTION:
Hyperglucagonemia is a common condition in obesity, prediabetes and type 2 diabetes. It increases the hepatic glucose production, thus contributing to type 2-diabetic hyperglycemia. In the current study we wish to examine whether non-alcoholic fatty disease (NAFLD) results in hepatic glucagon resistance. This could result in hyperglucagonemia through a feedback mechanism acting on the level of pancreatic alpha cells. Cirrhosis and type 1 diabetes, respectively, has previously been shown to be associated with hepatic glucagon resistance but it has not been examined in relation to NAFLD in humans so far.

ELIGIBILITY:
Inclusion Criteria:

* Normal fasting plasma glucose and HbA1c < 6.0%
* Between 18.5 and 25 kg/m2 or between 30 and 40 kg/m2
* Normal haemoglobin
* Normal coagulation factor II, VII and X, INR and thrombocytes
* Age above 25 years
* Informed consent

Exclusion Criteria:

* Diabetes
* Prediabetes (impaired glucose tolerance and/or impaired fasting plasma glucose)
* First-degree relatives with diabetes
* Nephropathy (eGFR < 60ml/min and/or albuminuria)
* Liver disease (ALAT and/or serum ASAT >2x normal values)
* Use of anticoagulative medicine like Clopidogrel og Warfarin
* Pregnancy and/or breastfeeding
* Age above 80 years
* Any condition that the investigator feels would interfere with trial participation

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Endogenous glucose production | 0-180 min
Amino acid metabolism | 0-180 min

SECONDARY OUTCOMES:
Degree of steatosis | baseline
Total RNA sequencing of liver biopsies | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Diabetes Research, Gentofte Municipality, Denmark

REFERENCES:
- [Background] Mitrakou A, Kelley D, Veneman T, Jenssen T, Pangburn T, Reilly J, Gerich J. Contribution of abnormal muscle and liver glucose metabolism to postprandial hyperglycemia in NIDDM. Diabetes. 1990 Nov;39(11):1381-90. doi: 10.2337/diab.39.11.1381. PMID 2121568
- [Background] Gromada J, Franklin I, Wollheim CB. Alpha-cells of the endocrine pancreas: 35 years of research but the enigma remains. Endocr Rev. 2007 Feb;28(1):84-116. doi: 10.1210/er.2006-0007. Epub 2007 Jan 16. PMID 17261637
- [Background] Knop FK, Aaboe K, Vilsboll T, Volund A, Holst JJ, Krarup T, Madsbad S. Impaired incretin effect and fasting hyperglucagonaemia characterizing type 2 diabetic subjects are early signs of dysmetabolism in obesity. Diabetes Obes Metab. 2012 Jun;14(6):500-10. doi: 10.1111/j.1463-1326.2011.01549.x. Epub 2012 Jan 17. PMID 22171657
- [Background] Faerch K, Pilgaard K, Knop FK, Hansen T, Pedersen O, Jorgensen T, Holst JJ. Incretin and pancreatic hormone secretion in Caucasian non-diabetic carriers of the TCF7L2 rs7903146 risk T allele. Diabetes Obes Metab. 2013 Jan;15(1):91-5. doi: 10.1111/j.1463-1326.2012.01675.x. Epub 2012 Sep 9. PMID 22862926
- [Background] Mitrakou A, Kelley D, Mokan M, Veneman T, Pangburn T, Reilly J, Gerich J. Role of reduced suppression of glucose production and diminished early insulin release in impaired glucose tolerance. N Engl J Med. 1992 Jan 2;326(1):22-9. doi: 10.1056/NEJM199201023260104. PMID 1727062
- [Background] Unger RH, Orci L. The essential role of glucagon in the pathogenesis of diabetes mellitus. Lancet. 1975 Jan 4;1(7897):14-6. doi: 10.1016/s0140-6736(75)92375-2. PMID 46337
- [Background] Liljenquist JE, Mueller GL, Cherrington AD, Keller U, Chiasson J-L, Perry JM, Lacy WW, Rabinowitz D. Evidence for an important role of glucagon in the regulation of hepatic glucose production in normal man. J Clin Invest. 1977 Feb;59(2):369-74. doi: 10.1172/JCI108649. PMID 833282
- [Background] Ferrannini E, Muscelli E, Natali A, Gabriel R, Mitrakou A, Flyvbjerg A, Golay A, Hojlund K; Relationship between Insulin Sensitivity and Cardiovascular Disease Risk (RISC) Project Investigators. Association of fasting glucagon and proinsulin concentrations with insulin resistance. Diabetologia. 2007 Nov;50(11):2342-7. doi: 10.1007/s00125-007-0806-x. Epub 2007 Sep 11. PMID 17846745
- [Background] Charbonneau A, Couturier K, Gauthier MS, Lavoie JM. Evidence of hepatic glucagon resistance associated with hepatic steatosis: reversal effect of training. Int J Sports Med. 2005 Jul-Aug;26(6):432-41. doi: 10.1055/s-2004-821225. PMID 16037884
- [Background] Longuet C, Robledo AM, Dean ED, Dai C, Ali S, McGuinness I, de Chavez V, Vuguin PM, Charron MJ, Powers AC, Drucker DJ. Liver-specific disruption of the murine glucagon receptor produces alpha-cell hyperplasia: evidence for a circulating alpha-cell growth factor. Diabetes. 2013 Apr;62(4):1196-205. doi: 10.2337/db11-1605. Epub 2012 Nov 16. PMID 23160527
- [Background] Bhathena SJ, Voyles NR, Smith S, Recant L. Decreased glucagon receptors in diabetic rat hepatocytes. Evidence for regulation of glucagon receptors by hyperglucagonemia. J Clin Invest. 1978 Jun;61(6):1488-97. doi: 10.1172/JCI109069. PMID 207737
- [Background] Kahn SE, Prigeon RL, McCulloch DK, Boyko EJ, Bergman RN, Schwartz MW, Neifing JL, Ward WK, Beard JC, Palmer JP, et al. Quantification of the relationship between insulin sensitivity and beta-cell function in human subjects. Evidence for a hyperbolic function. Diabetes. 1993 Nov;42(11):1663-72. doi: 10.2337/diab.42.11.1663. PMID 8405710
- [Background] Jimba S, Nakagami T, Takahashi M, Wakamatsu T, Hirota Y, Iwamoto Y, Wasada T. Prevalence of non-alcoholic fatty liver disease and its association with impaired glucose metabolism in Japanese adults. Diabet Med. 2005 Sep;22(9):1141-5. doi: 10.1111/j.1464-5491.2005.01582.x. PMID 16108839
- [Background] Gupte P, Amarapurkar D, Agal S, Baijal R, Kulshrestha P, Pramanik S, Patel N, Madan A, Amarapurkar A, Hafeezunnisa. Non-alcoholic steatohepatitis in type 2 diabetes mellitus. J Gastroenterol Hepatol. 2004 Aug;19(8):854-8. doi: 10.1111/j.1440-1746.2004.03312.x. PMID 15242486
- [Background] Akbar DH, Kawther AH. Nonalcoholic fatty liver disease in Saudi type 2 diabetic subjects attending a medical outpatient clinic: prevalence and general characteristics. Diabetes Care. 2003 Dec;26(12):3351-2. doi: 10.2337/diacare.26.12.3351-a. No abstract available. PMID 14633828
- [Background] Seghieri M, Rebelos E, Gastaldelli A, Astiarraga BD, Casolaro A, Barsotti E, Pocai A, Nauck M, Muscelli E, Ferrannini E. Direct effect of GLP-1 infusion on endogenous glucose production in humans. Diabetologia. 2013 Jan;56(1):156-61. doi: 10.1007/s00125-012-2738-3. Epub 2012 Oct 12. PMID 23064290
- [Background] Hare KJ, Vilsboll T, Asmar M, Deacon CF, Knop FK, Holst JJ. The glucagonostatic and insulinotropic effects of glucagon-like peptide 1 contribute equally to its glucose-lowering action. Diabetes. 2010 Jul;59(7):1765-70. doi: 10.2337/db09-1414. Epub 2010 Feb 11. PMID 20150286
- [Derived] Gilliam-Vigh H, Suppli MP, Heimburger SMN, Lund AB, Knop FK, Ellegaard AM. Cholesin mRNA Expression in Human Intestinal, Liver, and Adipose Tissues. Nutrients. 2025 Feb 8;17(4):619. doi: 10.3390/nu17040619. PMID 40004948
- [Derived] Suppli MP, Bagger JI, Lelouvier B, Broha A, Demant M, Konig MJ, Strandberg C, Lund A, Vilsboll T, Knop FK. Hepatic microbiome in healthy lean and obese humans. JHEP Rep. 2021 Apr 27;3(4):100299. doi: 10.1016/j.jhepr.2021.100299. eCollection 2021 Aug. PMID 34169247
- [Derived] Suppli MP, Bagger JI, Lund A, Demant M, van Hall G, Strandberg C, Konig MJ, Rigbolt K, Langhoff JL, Wewer Albrechtsen NJ, Holst JJ, Vilsboll T, Knop FK. Glucagon Resistance at the Level of Amino Acid Turnover in Obese Subjects With Hepatic Steatosis. Diabetes. 2020 Jun;69(6):1090-1099. doi: 10.2337/db19-0715. Epub 2020 Jan 23. PMID 31974144